CLINICAL TRIAL: NCT01569269
Title: A Randomized, Four-Arm Study Comparing Reiki, Yoga, Meditation, or Patient Education Group for Addressing Symptoms of Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Effects of Reiki, Yoga, Meditation, on the Physical and Psychological Symptoms of Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, Paul Clark, PhD, Assistant Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6870
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Peripheral Neuropathy
Keywords: chemotherapy induced peripheral neuropathy; cancer; psychological distress; mindfulness; complementary and alternative
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neoplasms | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Yoga (Experimental): See intervention description
  Interventions: Behavioral: Yoga Intervention
- Meditation (Experimental): See intervention description
  Interventions: Behavioral: Meditation Intervention
- Reiki (Experimental): see intervention description
  Interventions: Behavioral: Reiki
- Holistic Education (Active Comparator): see intervention description
  Interventions: Other: Holistic Education

INTERVENTIONS:
Behavioral: Yoga Intervention — The yoga intervention will take place for one hour per week for six weeks. All sessions will be guided by a Registered Yoga Teacher (RYT) who is also a Licensed Clinical Social Worker (LCSW).
  Each yoga session will follow a similar protocol. The introductory period (10 minutes) will focus participants on increasing interoceptive and proprioceptive capacity. The main segment is comprised of a series of yoga postures that progress from lying or seated postures that provide gentle muscle stretching to standing stretches that increase balance and flexibility. The postures will be introduced, practiced, and combined with breathing exercises for forty minutes.
  The conclusion of the session will be comprised of 10 minutes of relaxation.
  Arms: Yoga
Behavioral: Meditation Intervention — The meditation intervention will be conducted weekly for weeks. Each class will follow a similar protocol: During the one-hour meeting, participants will focus on developing attention to the breath. In a supine or seated position and with eyes closed, participants will be guided to attend solely to their breathing. As physical sensations, thoughts, and emotions begin to arise, participants will be taught to recognize, acknowledge, and accept the presence of the sensations or emotions and then to step back, release the thought or sensation, and refocus attention toward the breath At the conclusion of each meeting, the meditation instructor will encourage participants to voluntarily engage in daily meditation practices.
  Arms: Meditation
Behavioral: Reiki — The Reiki intervention will be conducted for one hour per week for 6 weeks. Protocol for each session: Briefly meet with the Reiki practitioner to review experiences with symptoms of CIPN. Then, the participant will be directed to lie supine and fully clothed on a massage table. Beginning at the top of the head, the practitioner will move inferiorly and pause while holding their hands above, but facing the participant at each energy point until reaching the feet. Upon reaching the participant's feet, the participant will roll from the supine position to a prone position and the process repeated. After being guided to a seated position on the massage table, the practitioner will spend a few moments in conversation with the participation before ending the session.
  Arms: Reiki
Other: Holistic Education — The psychoeducational intervention will be presented in a traditional classroom format with weekly one hour meetings taking place during the six week study period. Each class meeting will address specific aspects of CIPN. Participants will be presented with content related to basic neuroanatomy, physiology, the effects of chemotherapy on peripheral nervous system, how available allopathic treatments (pharmacological/psychopharmacological) can be helpful, and psychosocial issues related to CIPN. The final week of the psychoeducational group will include the identification of complementary interventions that may be of help to people living with CIPN.
  Arms: Holistic Education

SUMMARY:
The purpose of this study is to test whether people with symptoms of chemotherapy-induced peripheral neuropathy (CIPN) receive physical or psychological benefits from participating in a six-week Reiki, Yoga, Meditation, or Educational experience.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a side effect that occurs with many of the most common chemotherapeutic agents used to treat cancer. Typically, CIPN is experienced as tingling, burning, numbness, or pain in the upper and lower extremities and other parts of the body. Severity of symptoms can range from bothersome to disabling and can have profoundly negative effects on quality of life. Although the specific incidence or prevalence of CIPN is unknown, it is generally estimated at 30 to 40 percent in patients who have received the classes of chemotherapeutic agents used to treat breast, colon, and lung, cancers, and lymphomas. There are no treatments or drugs that consistently ameliorate or lead to the reversal of CIPN symptoms.Typically, symptoms of CIPN are considered along with other pain symptoms and treated with opioids and analgesics. Additionally, the prescription of anticonvulsant medications and tricyclic antidepressants can help alleviate neuropathic pain. While these strategies can provide relief from cancer-related pain, they often yield limited results for symptoms of CIPN. With few allopathic treatment alternatives for attenuating the symptoms of CIPN, people living with these symptoms have few options other than to endure them.

Unlike treatments based upon nociceptive and neuropathic models of pain that regard the pain response as the outcome of a finite and mechanistic chain of biochemical events, complementary treatments acknowledge the interpenetrating nature of the relationships between body, mind, and spirit. Typically, complementary or integrative health strategies incorporate psychological, emotional, and spiritual elements along with biochemical strategies when addressing pain. Of particular interest in the proposed pilot study are complementary techniques that include Yoga, Meditation, and Reiki.

Utilizing a pretest-posttest control group design with random assignment, this four-arm experimental pilot study will be undertaken to determine the feasibility of three complementary approaches in reducing the signs and symptoms of CIPN. This design was chosen for its ability to support causal inference while managing threats to internal and external design validity. The use of random assignment in the development of intervention and comparison groups will strengthen the ability of this design to manage threats to internal validity more efficiently. This pilot study involves the collection of quantitative data from self-administered instruments that have been designed to measure health related quality of life, symptoms of neurotoxicity, psychological distress, and mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* participants must be of at least 18 years of age,
* participants must have persistent symptoms of CIPN resulting from treatment with vinca alkaloid, taxane, platinum class chemotherapies or immunomodulators (Thalidomide) or antineoplastic agents (Velcade) for a known cancer diagnosis
* participants must have completed chemotherapy at least three months prior to beginning the study,
* participants cannot concurrently receive chemotherapy treatment for cancer, nor
* actively take part in one of the complementary modalities offered in this pilot study.
* participants will be required to have an ability to comfortably speak, read, and understand English.
* participants must be fully oriented and possess the capacity to understand and provide informed consent for participation in the study.

Exclusion Criteria:

* failure to meet any one of the inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
FACT GOG-ntx scale | change from baseline in quality of life and symptoms of neurotoxicity in 6 weeks
  This scale measures two outcomes:symptoms of neurotoxicity and quality of life. The FACT GOG-ntx combines the 27-item general Functional Assessment of Cancer Therapy scale (FACT-G) with an 11-item neurotoxicity subscale. Completion of the FACT-G does not require assistance and can be completed in less than five minutes. Cronbach's coefficient for each item on this scale has been demonstrated at 0.70 or higher, and the instrument is sensitive to respondent changes over time.

SECONDARY OUTCOMES:
The Brief Symptom Inventory - 18 (BSI-18) | change from baseline in quality of life and symptoms of neurotoxicity in 6 weeks
  The BSI-18 is an 18-item brief psychological screening instrument that has been designed to measure distress and yields a global distress score as well as subscale scores for somatic concerns, anxiety, and depression. The BSI-18 has been found to have good internal reliability with a Cronbach's alpha value of 0.89
Mindful Attention Awareness scale (MAAS) | change from baseline in quality of life and symptoms of neurotoxicity in 6 weeks
  The MAAS is a 15-item scale that is self-administered, requires no assistance to complete, and can be taken in five minutes or less. The instrument was developed to evaluate states of mindfulness or the respondent's capacity to simply observe and be aware of internal and external events in the present moment as a method of self-regulation. Internal reliability of items on the MAAS has been established with Cronbach's Alpha coefficients at 0.80 or higher per item.

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Clark, PhD, Principal Investigator — George Mason University
Locations (1):
- Life with Cancer Family Center, Fairfax, Virginia, United States